CLINICAL TRIAL: NCT04127513
Title: Comparison of Efficacy and Safety Between Moisturising Cream Containing 12% Ammonium Lactate AND 10% Urea in Geriatric With Xerosis Cutis: Double Blind Randomised Controlled Trial
Brief Title: Comparison of 12% Ammonium Lactate and 10% Urea Cream in Geriatric With Xerosis Cutis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Eyleny Meisyah Fitri, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ThesisEyleny
Record Dates: First submitted 2019-10-10; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Xerosis Cutis
Keywords: xerosis cutis; geriatric; 12% ammonium lactate; 10% urea
MeSH Terms: interventions — Lactic Acid; Urea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: same vehicle base ingredients, colour, smell, and packaging
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 12% AMMONIUM LACTATE (Experimental): Matching paired subject was conducted on 40 residents. Test subject received two different randomized moisturizing creams to be applied on two separate locations on the lower limbs twice a day for 4 weeks. One of the moisturising cream contained active ingredient 12% ammonium lactate. The evaluation of specified symptom sum score (SRRC), skin capacitance (SCap), transepidermal water loss (TEWL), and side effects were measured at baseline, week-2 and week-4 after therapy, and week-5 one week after therapy cessation.
  Interventions: Drug: Ammonium Lactate
- 10% UREA (Active Comparator): Matching paired subject was conducted on 40 residents. Test subject received two different randomized moisturizing creams to be applied on two separate locations on the lower limbs twice a day for 4 weeks. One of the moisturising cream contained active ingredient 10% urea. The evaluation of specified symptom sum score (SRRC), skin capacitance (SCap), transepidermal water loss (TEWL), and side effects were measured at baseline, week-2 and week-4 after therapy, and week-5 one week after therapy cessation.
  Interventions: Drug: Urea

INTERVENTIONS:
Drug: Ammonium Lactate — 12% ammonium lactate moisturizing cream
  Arms: 12% AMMONIUM LACTATE
Drug: Urea — 10% urea moisturizing cream
  Arms: 10% UREA

SUMMARY:
This study aims to compare the efficacy and safety between moisturizing cream containing 12% ammonium lactate and 10% urea in geriatric with xerosis cutis. A double-blind randomized controlled trial with matching paired subject was conducted on 40 residents of a nursing home in Jakarta. Specified symptom sum score (SRRC), skin capacitance (SCap), transepidermal water loss (TEWL), and side effects were measured at baseline, week-2 and week-4 after therapy, and week-5 one week after therapy cessation. After a week of preconditioning, each subject received two different moisturizing creams to be applied on separate lower limbs.

DETAILED DESCRIPTION:
Dry skin or xerosis cutis is widely known skin health issue in geriatric population with prevalence rate ranges between 29.5 - 85.5%. One of the internal etiological factors is decreased production of natural moisturizing factor as a humectant. Application of moisturizer is the mainstay treatment. Moisturizer with humectant property, like lactate and urea, could restore skin hydration and barrier dysfunction. This study aims to compare the efficacy and safety between moisturizing cream containing 12% ammonium lactate and 10% urea in geriatric with xerosis cutis.

ELIGIBILITY:
Inclusion Criteria:

* presenting with clinical diagnosis of xerosis cutis or with using the specified symptom sum score (SRRC)
* able to communicate well and perform daily activities independently
* willing to follow the research and sign the informed consent

Exclusion Criteria:

* sensitive to the ingredients in the formulations
* suffer from dermatitis or skin inflammation at the test site
* erythema and fissure values based on SRRC value >2

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
First Evaluation of Specified Symptom Sum Score (SRRC) | initial visit (day 1)
  System with grading of scaliness, roughness, redness, and cracks with score ranges from 0-12 because the redness and cracks scores were limited to 2. Performed before therapy.
Second Evaluation of Specified Symptom Sum Score (SRRC) | Change of SSRC at day 15 from initial visit
  System with grading of scaliness, roughness, redness, and cracks with score ranges from 0-12 because the redness and cracks scores were limited to 2. Performed during therapy.
Third Evaluation of Specified Symptom Sum Score (SRRC) | Change of SSRC at day 29 from initial visit
  System with grading of scaliness, roughness, redness, and cracks with score ranges from 0-12 because the redness and cracks scores were limited to 2. Performed during therapy.
Fourth Evaluation of Specified Symptom Sum Score (SRRC) | Change of SSRC at day 36
  System with grading of scaliness, roughness, redness, and cracks with score ranges from 0-12 because the redness and cracks scores were limited to 2. Performed after 1 week of therapy discontinuation
First Evaluation of Skin Capacitance (SCap) | Performed at initial visit (day-1)
  Assess the skin barrier homeostasis condition using Corneometer® CM 825 (Courage - Khazaka, Germany). Performed before therapy.
Second Evaluation of Skin Capacitance (SCap) | Change of SCap at day-15
  Assess the skin barrier homeostasis condition using Corneometer® CM 825 (Courage - Khazaka, Germany). Performed during therapy.
Third Evaluation of Skin Capacitance (SCap) | Change of SCap at day-29
  Assess the skin barrier homeostasis condition using Corneometer® CM 825 (Courage - Khazaka, Germany). Performed during therapy.
Fourth Evaluation of Skin Capacitance (SCap) | Change of SCap at day-36
  Assess the skin barrier homeostasis condition using Corneometer® CM 825 (Courage - Khazaka, Germany). Performed after 1 week of therapy discontinuation
First Evaluation of Transepidermal Water Loss (TEWL) | Performed at initial visit (day-1)
  Assess the skin barrier homeostasis condition using Tewameter® TM300 before therapy.
Second Evaluation of Transepidermal Water Loss (TEWL) | Change of TEWL at day-15 from initial visit
  Assess the skin barrier homeostasis condition using Tewameter® TM300. Performed during therapy.
Third Evaluation of Transepidermal Water Loss (TEWL) | Change of TEWL at day-29 from initial visit
  Assess the skin barrier homeostasis condition using Tewameter® TM300. Performed during therapy.
Fourth Evaluation of Transepidermal Water Loss (TEWL) | Change of TEWL at day-36 from initial visit
  Assess the skin barrier homeostasis condition using Tewameter® TM300. Performed after 1 week of therapy discontinuation.
First Side Effect Evaluation | Performed at 2 weeks after therapy (day-15)
  Subjective by the presence of contact dermatitis, folliculitis, and miliaria; objective by complaints of pruritus, sore, or stinging.
Second Side Effect Evaluation | Performed at day-29 (4 weeks after therapy)
  Subjective by the presence of contact dermatitis, folliculitis, and miliaria; objective by complaints of pruritus, sore, or stinging.
Third Side Effect Evaluation | Performed at day-36 (5 weeks after therapy)
  Subjective by the presence of contact dermatitis, folliculitis, and miliaria; objective by complaints of pruritus, sore, or stinging. Performed after 1 week of therapy discontinuation

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine University of Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No